CLINICAL TRIAL: NCT04483609
Title: SF-QUALIVEEN Turkish Cultural Adaptation, Validity and Reliability Study
Brief Title: SF-QUALIVEEN Turkish Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Uğur OVACIK, Instructor, Istanbul Aydın University
Other Study IDs: 2018/23-21
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; urological dysfunction; assessment; scale
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-test Group: 10 people with multiple sclerosis. The eligibility criteria were: (1) age 18-65; (2) definitive diagnosis of MS according to McDonald criteria; (3) ability to read and write in Turkish. The exclusion criteria are: (1) acute attacks of MS (within 3 months); (2) cognitive impairment (Mini Mental test result 24 points and below); (3) any chronic disease other than MS; (4) active malignant tumors; (5) symptomatic urinary tract infections; (6) patients who changed treatment within the test-retest period.
  Interventions: Other: Questionnaire administration pre test
- Validation and Reliability Group: 80 people with multiple sclerosis. The eligibility criteria were: (1) age 18-65; (2) definitive diagnosis of MS according to McDonald criteria; (3) ability to read and write in Turkish. The exclusion criteria are: (1) acute attacks of MS (within 3 months); (2) cognitive impairment (Mini Mental test result 24 points and below); (3) any chronic disease other than MS; (4) active malignant tumors; (5) symptomatic urinary tract infections; (6) patients who changed treatment within the test-retest period.
  Interventions: Other: Questionnaire administration validation and reliability

INTERVENTIONS:
Other: Questionnaire administration pre test — After the translation and cultural adaptation of the SF-Qualiveen scale is completed, face-to-face pre-test will be performed on 10 patients with multiple sclerosis.
  Groups: pre-test Group
Other: Questionnaire administration validation and reliability — After the pre-test is completed, if necessary, arrangements will be made, and then the validity and reliability of SF-Qualiveen will be made in 80 individuals with Multiple Sclerosis.First of all, participants will be asked to complete two questionnaires (SF-Qualiveen and Urinary Distress Inventory). Two weeks after this assessment, they will be asked to respond to SF-Qualiveen again.
  Groups: Validation and Reliability Group

SUMMARY:
Urological dysfunction is common in patients with Multiple Sclerosis (MS) and its prevalence has been reported at a high rate of 32-97%. Bladder dysfunction is associated with a significant deterioration in the quality of life of people with MS. In chronic diseases such as MS, patients experiences need to be measured directly in order to have information about patients perceptions about the effect of the disease on quality of life. However, there are a small number of valid and reliable Turkish scales on this subject.SF-Qualiveen is a validated scale for patients with MS who assess the urinary-specific quality of life by examining the impact of a wide range of bladder problems.The aim of our study is to make the Turkish cultural adaptation, validity and reliability of the SF-Qualiveen scale.

DETAILED DESCRIPTION:
The aim of this study is to reveal the Turkish cultural adaptation, validity and reliability of the SF-Qualiveen scale. In our study, Sf-Qualiveen and Urogenital Distress Inventory (UDI-6) scales will be used. Pre-testing will be done in 10 patients with multiple sclerosis.Then, the validity and reliability of the scale will be performed in 80 patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65;
2. definitive diagnosis of MS according to McDonald criteria;
3. ability to read and write in Turkish.

Exclusion Criteria:

1. acute attacks of MS (within 3 months);
2. cognitive impairment (Mini Mental test result 24 points and below);
3. any chronic disease other than MS;
4. active malignant tumors;
5. symptomatic urinary tract infections;
6. patients who changed treatment within the test-retest period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-test: 10 patients with multiple sclerosis will be evaluated.Inclusion and exlusion criteria listed above.
  Validation and reliability: 70 patients with multiple sclerosis will be evaluated.Inclusion and exlusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
SF-Qualiveen score | Baseline
  To evaluate the impact of urological problems on quality of life

SECONDARY OUTCOMES:
Urogenital Distress Inventory (UDI-6) | Baseline
  To assess problems caused by urinary symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided